CLINICAL TRIAL: NCT00644163
Title: NIMH Multisite HIV/STD Prevention Trial for African American Couples
Brief Title: Effectiveness of a Risk Reduction Program in Preventing the Transmission of HIV and Sexually Transmitted Diseases in African-American Couples
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH); University of California, Los Angeles (Other); Emory University (Other); Columbia University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Purpose: Prevention
Other Study IDs: U10MH078819 (NIH); U10MH078819 (NIH); DAHBR 9A-ASGT
Record Dates: First submitted 2008-03-24; First posted 2008-03-26 (Estimated); Last update posted 2014-01-27 (Estimated); Status verified 2009-02

CONDITIONS: HIV Infections; Sexually Transmitted Disease
Keywords: HIV; STI; Risk Reduction; Couples; African American; HIV Seronegativity
MeSH Terms: conditions — HIV Infections; Sexually Transmitted Diseases; Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive Eban HIV/STD Risk Reduction Intervention.
  Interventions: Behavioral: Eban HIV/STD Risk Reduction Intervention
- 2 (Active Comparator): Participants will receive Eban Health Promotion Intervention.
  Interventions: Behavioral: Eban Health Promotion Intervention

INTERVENTIONS:
Behavioral: Eban HIV/STD Risk Reduction Intervention — The eight-session Eban HIV/STD Risk Reduction Intervention is embedded in a cultural context and is gender tailored in its prevention messages and activities. Sessions will focus on the couple and will teach the couple about communication skills. The approach will draw upon social cognitive theory, an ecological framework, and HIV/STD risk-reduction research with inner-city African-American populations.
  Arms: 1
Behavioral: Eban Health Promotion Intervention — The eight-session Eban Health Promotion Intervention is guided by a social cognitive approach that engages health promotion skills. Sessions will focus on the individual and will provide factual information on health, screening, exercise, diet management, and medication adherence.
  Arms: 2

SUMMARY:
This study will evaluate the effectiveness of a risk-reduction program in preventing the transmission of HIV and sexually transmitted diseases among African-American heterosexual couples, with one partner having been previously diagnosed with an HIV infection.

DETAILED DESCRIPTION:
The transmission of sexually transmitted diseases (STDs), including HIV, is a major public health concern, especially among minority groups in the United States. Although STDs are prevalent across all racial and ethnic groups in the United States, the rate of STD infection is disproportionately higher for African Americans than for white Americans. African Americans have higher rates of HIV, chlamydia, gonorrhea, syphilis, and herpes than white Americans. An important part of the prevention process is early education on HIV to reduce sexual-risk behavior and to promote safe sexual practices. Interventions are needed in a variety of settings to extensively address African Americans' risk of STDs, including HIV. Although most HIV/STD risk-reduction interventions are conducted at the individual level, a couple-based approach may be more effective and consistent with cultural values. This study will compare the effectiveness of the Eban HIV/STD Risk Reduction Intervention with the Eban Health Promotion Intervention in reducing the risk of STDs among African-American HIV-serodiscordant heterosexual couples.

Participation in this study will last 12 months. All participants will first undergo baseline assessments that will consist of questionnaires and biospecimen collection for STD testing. Participants will then be assigned randomly to one of two treatment groups: the Eban HIV/STD Risk Reduction Intervention group or the Eban Health Promotion Intervention group. Both groups will participate in weekly 2-hour sessions over 8 weeks. The sessions will include couple and group sessions led by trained male and female co-facilitators. The Eban HIV/STD Risk Reduction Intervention sessions will focus on the couple and will teach the couple about communication skills. The approach will draw upon social cognitive theory, an ecological framework, and HIV/STD risk-reduction research with inner-city African-American populations. The Eban Health Promotion Intervention sessions will focus on the individual and will provide factual information on health, screening, exercise, diet management, and medication adherence. Follow-up visits for all participants will occur at Months 3, 6, and 12 and will include repeat baseline assessments.

ELIGIBILITY:
Inclusion Criteria:

* Each partner agrees that the relationship has lasted at least 6 months before study entry
* Each partner intends to remain together for at least 12 months after study entry (e.g., state independently that he/she is confident or very confident that they will remain together)
* At least one partner of the couple reports having unprotected intercourse at least once in the 90 days before study entry
* Neither partner has plans to relocate beyond a reasonable distance from the study site
* At least one partner is African American
* At least one partner agrees that he/she is not planning pregnancy within the next 18 months after study entry
* Each partner is aware of his/her partner's HIV serostatus
* Only one partner is HIV seropositive and has known his or her status for at least 3 months before study entry

Exclusion Criteria:

* One or both partners do not have an address where they can receive mail
* One or both partners have significant psychiatric, physical, or neurological impairment that would limit their effective participation as confirmed on a Mini Mental State Examination and/or Quick Test
* History of severe physical or sexual abuse in the 1 year before study entry in the current relationship (e.g., significant enough to require medical, psychological, and/or legal intervention)
* One or both partners are unwilling or unable to commit to participate in the study through to completion
* Both partners have previously participated in an HIV sexual risk-reduction intervention for couples in the 12 months before study entry
* One or both partners are not fluent in English as determined by the informed consent process

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1070 (Actual)
Dates: Start 2003-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
Self-reported proportion of condom-protected sexual intercourse | Measured at Month 12
Occurrence of STDs (chlamydia, gonorrhea, and trichomonas) | Measured at Month 12

SECONDARY OUTCOMES:
Unprotected sex occurrence | Measured at Month 12
Number of sexual partners | Measured at Month 12

CONTACTS AND LOCATIONS:
Overall Officials: John Jemmott, PhD, Principal Investigator — University of Pennsylvania; Nabila el-Bassel, DSW, Principal Investigator — Columbia University; Gail Wyatt, PhD, Principal Investigator — University of California, Los Angeles; Gina Wingood, ScD, Principal Investigator — Emory University; J. Richard Landis, PhD, Principal Investigator — University of Pennsylvania/Data Coordinating Center
Locations (4):
- United States (4):
  - UCLA, Los Angeles, California
  - Emory University, Atlanta, Georgia
  - Columbia University, New York, New York
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Derived] Hamilton AB, Mittman BS, Williams JK, Liu HH, Eccles AM, Hutchinson CS, Wyatt GE. Community-based implementation and effectiveness in a randomized trial of a risk reduction intervention for HIV-serodiscordant couples: study protocol. Implement Sci. 2014 Jun 20;9:79. doi: 10.1186/1748-5908-9-79. PMID 24950708
- [Derived] El-Bassel N, Jemmott JB 3rd, Landis JR, Pequegnat W, Wingood GM, Wyatt GE, Bellamy SL; National Institute of Mental Health Multisite HIV/STD Prevention Trial for African-American Couples Group. Intervention to influence behaviors linked to risk of chronic diseases: a multisite randomized controlled trial with African-American HIV-serodiscordant heterosexual couples. Arch Intern Med. 2011 Apr 25;171(8):728-36. doi: 10.1001/archinternmed.2011.136. PMID 21518939
- [Derived] El-Bassel N, Jemmott JB, Landis JR, Pequegnat W, Wingood GM, Wyatt GE, Bellamy SL; NIMH Multisite HIV/STD Prevention Trial for African American Couples Group. National Institute of Mental Health Multisite Eban HIV/STD Prevention Intervention for African American HIV Serodiscordant Couples: a cluster randomized trial. Arch Intern Med. 2010 Sep 27;170(17):1594-601. doi: 10.1001/archinternmed.2010.261. Epub 2010 Jul 12. PMID 20625011